CLINICAL TRIAL: NCT05495282
Title: Traditional Lecture Versus Procedural Video Randomized Trial: Comparative Analysis of Instructional Methods for Teaching Baclofen Pump Management
Brief Title: Traditional Lecture Versus Procedural Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-21-1513
Record Dates: First submitted 2022-08-05; First posted 2022-08-10 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Educational Problems

STUDY DESIGN:
Intervention Model Description: Single-center cross over design
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assessor will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Traditonal Lecture (No Intervention): Group A (n=30) will receive a baclofen pump refill and programming instruction via the traditional lecture method performed by a single faculty member. The traditional lecture will consist of a PowerPoint lecture for 30 minutes, a demonstration of the refilling and programming technique for 10 minutes, and participant hands-on practice refilling and programming a baclofen pump for 20 minutes. Group A will have time to practice refilling and programming baclofen pumps with the guidance of a single faculty member during the traditional 60-minute lecture.
- Group B: Microvideo (Experimental): Group B (n=30) will receive an asynchronous 10-minute micro-video on the topic for which no face-to-face interaction with faculty will be conducted. The micro-video will be provided on a 12.9-inch iPad pro for each participant to view individually. The micro-video group will also have the opportunity to practice pump refilling before the post-evaluation. Participants in Group B will have the micro-video instruction available while practicing hands-on baclofen pump refilling and programming. The maximum time allowed to view the micro-video and practice hands-on baclofen pump refilling and programming will be 30-minutes. The time that each participant in group B spends reviewing the micro-video and practicing hands-on pump refilling and programming will be recorded. The participant may view and rewind the video as many times as needed in the 30-minute period. The live demonstration and the procedural video describe identical steps involved in refilling and programming the baclofen pump.
  Interventions: Other: Microvideo

INTERVENTIONS:
Other: Microvideo — Asynchronous 10-minute micro-video on the topic for which no face-to-face interaction with faculty will be conducted.
  Arms: Group B: Microvideo

SUMMARY:
The study would consist of teaching pain management and physical medicine and rehabilitation physicians how to program and refill a baclofen pump with two different methods. A baclofen pump is a device that delivers a medication called baclofen to the spinal canal. The baclofen pump is surgically implanted near the abdomen, with a thin, flexible tube running to the spinal canal to deliver the medication. The study aims to measure the effectiveness of procedural video compared to traditional lectures in transferring skills for refilling and programming a baclofen pump. This will be a controlled study consisting of two randomly assigned groups of physicians with inexperience with refilling and programming baclofen pumps. Before randomization, all participants will be tested on baclofen pump refilling and programming on the baclofen pump simulator. The control group will then receive a traditional 60-minute lecture on teaching baclofen pump management, while the intervention group will watch a 10-minute video on baclofen pump management. The traditional lecture will consist of a PowerPoint lecture for 30 minutes, a demonstration of the refilling and programming technique for 10 minutes, and participant hands-on practice refilling and programming a baclofen pump for 20 minutes. The intervention group will have 30 minutes to view the video and practice hands-on baclofen pump refilling and programming. The video may be viewed as many times as needed over the 30 minutes. The participants will then be re-tested on baclofen pump refilling and programming on the simulator. Six to eight weeks later, the participants will have repeat testing on baclofen pump refilling and programming on the simulator to see if knowledge was retained over time. Once repeat testing is complete, the control group will review the 10-minute video, and the intervention group will receive the 60-minute traditional lecture. The study will conclude with an approximately 30-minute focus group discussing the two education methods.

DETAILED DESCRIPTION:
Day 1 - 6 to 8 hours:

The study will be performed at Carilion Roanoke Community Hospital. Participants will be enrolled in a study to evaluate traditional lecture versus an asynchronous micro-video for teaching baclofen pump refilling and programming skills. Demographic information will be collected for each participant (table 1). Six education sessions will be conducted with ten participants per session. The duration of the session will be six to eight hours. All participants will perform pre-intervention baclofen pump refilling and programming in the simulated environment graded using a rubric for baclofen pump management. A SynchroMed II baclofen pump simulator will be used to simulate baclofen pump refilling and programming during the study. The participant will interrogate the pump, refill the pump with simulated intrathecal baclofen, and program the pump by increasing the daily rate of intrathecal baclofen by 10%. The scenarios used for the study will be the same for all simulations. Subjects will be tested individually to eliminate any group practice effects of observing other subjects testing. The rubric will be graded and recorded by one consistent investigator. The rubric has a minimum score of 0.5 and a maximum score of 10, with four steps referred to as "fatal flaws" that must be completed correctly to receive a passing score. A passing score on the rubric is a 9/10 with no "fatal flaws." The rubric for baclofen pump management has been studied in physical medicine & rehabilitation residents, and non-published data showed a mean evaluation score and experience refilling and programming baclofen pumps to be highly correlated (Pearson coefficient = 0.899, p-value = 0.0489). Cronbach's alpha was calculated and was 0.91 showing good internal consistency.

Participants will be randomly allocated to either the micro-video intervention group or the traditional lecture control group. Randomization would be done using the random number generator formula in Microsoft Excel. They would be informed of their group allocation. The participants will not be blinded as they would come to know if they are placed in the intervention or the control group. Group A (n=30) will receive a baclofen pump refill and programming instruction via the traditional lecture method performed by a single faculty member. The traditional lecture will consist of a PowerPoint lecture for 30 minutes, a demonstration of the refilling and programming technique for 10 minutes, and participant hands-on practice refilling and programming a baclofen pump for 20 minutes. Group A will have time to practice refilling and programming baclofen pumps with the guidance of a single faculty member during the traditional 60-minute lecture. In contrast, Group B (n=30) will receive an asynchronous 10-minute micro-video on the topic for which no face-to-face interaction with faculty will be conducted. The micro-video will be provided on a 12.9-inch iPad pro for each participant to view individually. The micro-video group will also have the opportunity to practice pump refilling before the post-evaluation. Participants in Group B will have the micro-video instruction available while practicing hands-on baclofen pump refilling and programming. The maximum time allowed to view the micro-video and practice hands-on baclofen pump refilling and programming will be 30-minutes. The time that each participant in group B spends reviewing the micro-video and practicing hands-on pump refilling and programming will be recorded. The participant may view and rewind the video as many times as needed in the 30-minute period. The live demonstration and the procedural video describe identical steps involved in refilling and programming the baclofen pump.

The participants from both groups will then be subjected to post-intervention baclofen pump refilling and programming graded with the same rubric following exposure to the traditional lecture or asynchronous micro-video. The investigator that provided initial pre-intervention baclofen pump rubric grading will assess baclofen refilling and programming for both groups according to pre-specified criteria in the rubric. The investigator providing evaluation will be blinded to the instructional method. Subjects will be tested individually to eliminate any group practice effects of observing other subjects while testing. Rubric scoring will be recorded for both groups.

Day 2 - 4 to 5 hour:

Between six and eight weeks after the initial intervention, participants from both groups will perform a second post-intervention baclofen pump refilling and programming on a simulated patient with the same blinded investigator during six sessions of ten subjects each. This session will occur at Carilion Roanoke Community Hospital and will last four to five hours. Participants will be graded with the same rubric to see if knowledge was retained. Rubric scoring will be recorded for both groups. Subjects will be tested individually to eliminate any group practice effects of observing other subjects while testing. A traditional 60-minute lecture for Group B will follow the second post-intervention baclofen pump refilling and programming, and the asynchronous micro-video will be shared with Group A.

Following exposure to both methods of instruction, participants will provide feedback on the learning methods using structured focus groups (figure 1). Six focus group sessions will be performed with the ten subjects in each education session. Each focus group will last about 30 minutes to minimize participants' fatigue. One of the study investigators will serve as a trained moderator will lead the qualitative, semi-structured group interview to assess their overall experiences with traditional lecture versus an asynchronous micro-video (Appendix B). This will include new information learned by participants during the study, including discussing participant learning preferences that may inform future education practice for filling and programming baclofen pumps. The focus groups will be recorded and transcribed verbatim.

ELIGIBILITY:
Inclusion Criteria:

* Board Certified or Board Eligible in Physical Medicine & Rehabilitation or Pain Management
* A 25 to 70-year-old novice baclofen pump provider which is defined as refilling and programming less than ten baclofen pumps in simulation or clinical encounters in the past two years.

Exclusion Criteria:

* A experienced baclofen provider as defined refilling and programming more than ten baclofen pumps in simulation or clinical encounters in the past two years.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-06 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Rubric scores | 3 months
  The primary outcome of the proposed study is to measure the effectiveness of procedural micro-video compared to traditional lectures in transferring skills for refilling and programming a baclofen pump using the rubric for baclofen pump refilling and programming at three-time points (pre-intervention, post-intervention, and six to eight weeks following intervention).

SECONDARY OUTCOMES:
Perceived effectiveness of learning modality | 3 months
  The secondary learning outcome measures the learner's perceived effectiveness of procedural video compared with a traditional lecture using qualitative research methods.

CONTACTS AND LOCATIONS:
Overall Officials: Justin L Weppner, DO, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Roanoke Community Hospital, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weppner J, Conti A, Locklear TM, Mayer RS. Traditional Lecture Versus Procedural Video Randomized Trial: Comparative Analysis of Instructional Methods for Teaching Baclofen Pump Management. Am J Phys Med Rehabil. 2024 Jun 1;103(6):510-517. doi: 10.1097/PHM.0000000000002397. Epub 2023 Dec 21. PMID 38261785